CLINICAL TRIAL: NCT04913350
Title: Effect of Russian Current on Contralateral Muscle Strength in Adolescents Athlete :A Randomized Controlled Trial
Brief Title: Contralateral Effects of Russian Current on Adolescent Athlete
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Samah Mahmoud Sheha, principal investigator, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUS PT 012
Record Dates: First submitted 2021-04-03; First posted 2021-06-04 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Treatment Side Effects
Keywords: Tennis Elbow; Cross-Training; Electrical Stimulation
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Russian current and elbow support group (Experimental): participants in the experimental group will apply elbow support and will receive Russian current on biceps and triceps muscles of the unaffected elbow three therapy sessions per week for 4 weeks.
  Interventions: Other: Russian current; Device: elbow support
- elbow support group (Active Comparator): Participants in this group will apply elbow support only.
  Interventions: Device: elbow support

INTERVENTIONS:
Other: Russian current — One of the preferred common neuromuscular electrical stimulation techniques for muscle strengthening is the Russian current (RC) It stimulates almost all muscle motor units to contract synchronously, resulting in a greater muscle hypertrophy.
  Arms: Russian current and elbow support group
Device: elbow support — tennis elbow brace is recommended to decrease pain and improve function by restricting the movement of the forearm or relieving loads on the origin of the muscles of the extensor

SUMMARY:
The strength loss associated with immobilization causes long term decreases in performance and loss of hours of participation for athletes during rehabilitation period to regain a competitive form. Therefore, reducing such effects throughout the immobilization period is highly preferable. Cross-educational strength transfer to the inactive muscle by means of unilateral strength training may provide an opportunity to avoid strength loss and atrophy.

DETAILED DESCRIPTION:
After injury and/or surgery, neuromuscular electrical stimulation is widely used to train muscles and enhance muscle strength. and some studies have found it to be superior to voluntary exercise after immobilization . One of the preferred common NMES techniques for muscle strengthening is the Russian current (RC) It stimulates almost all muscle motor units to contract synchronously, resulting in a greater muscle hypertrophy. While some studies exist to confirm the efficacy of this current in the Russian language, there is very little evidence to support its use in English literature. The aim of our study is to investigate the effectiveness of cross education of Russian current on the strength of the contralateral inactive biceps and triceps muscles of the affected elbow in pediatrics athletes to decrease some of the negative effects of immobilization on muscle tissue and enhance recovery.

ELIGIBILITY:
Inclusion Criteria:

* 1 year experience in tennis training
* diagnosis of tennis elbow

Exclusion Criteria:

* Any contraindication to the application of electrotherapy
* upper limb surgery

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
muscle strength | 4 weeks
  The concentric isokinetic elbow flexors and extensors peak torque in Newton-meters, for the dominant side (affected side) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Samah M Sheha, PhD, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Misr university for science and technology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hendy AM, Spittle M, Kidgell DJ. Cross education and immobilisation: mechanisms and implications for injury rehabilitation. J Sci Med Sport. 2012 Mar;15(2):94-101. doi: 10.1016/j.jsams.2011.07.007. Epub 2011 Sep 15. PMID 21924681
- [Background] Wilkinson SB, Tarnopolsky MA, Grant EJ, Correia CE, Phillips SM. Hypertrophy with unilateral resistance exercise occurs without increases in endogenous anabolic hormone concentration. Eur J Appl Physiol. 2006 Dec;98(6):546-55. doi: 10.1007/s00421-006-0300-z. Epub 2006 Sep 14. PMID 16972050
- [Background] Akinoglu B, Kocahan T. Russian current versus high voltage current with isokinetic training on the quadriceps muscle strength and endurance. J Exerc Rehabil. 2020 Jun 30;16(3):272-278. doi: 10.12965/jer.2040260.130. eCollection 2020 Jun. PMID 32724785
- [Background] Ganesh GS, Kumari R, Pattnaik M, Mohanty P, Mishra C, Kaur P, Dakshinamoorthy A. Effectiveness of Faradic and Russian currents on plantar flexor muscle spasticity, ankle motor recovery, and functional gait in stroke patients. Physiother Res Int. 2018 Apr;23(2):e1705. doi: 10.1002/pri.1705. Epub 2018 Feb 8. PMID 29417699

DOCUMENTS (1):
  • Informed Consent Form (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04913350/ICF_000.pdf